CLINICAL TRIAL: NCT04154033
Title: Treatment of Chronic Itch in Atopic Dermatitis With Topical Naltrexone as Well as the Influence of Circadian Rhythm
Brief Title: Treatment of Chronic Itch in Atopic Dermatitis With Topical Naltrexone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DERM-2019-27870
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis; Pruritus; Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Dermatitis | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Circadian Rhythm of Itch (No Intervention): For the study arm A, to evaluate circadian rhythm of itching, patients will record for 7 days 6 times daily in a booklet the itch intensity on a visual analog scale (VAS) scale. These time points for itch intensity recording will be hours after time of awakening (AW), so they will be AW+2h, AW+4h, AW+6h, AW+8h, AW+10h, AW+12h. Patients are to document all their pruritus attacks at these time points. On day 8 the investigators will collect suction blisters (4-5 10mm blisters) at these 6 time points from unaffected skin on the trunk. For this purpose, the investigators will use the commercially available 47mm orifice plate (Electronic Diversities, Finksburg MD, USA) with 4-5 x10mm openings for each time point and use the 4-5 1mm blister roofs for harvesting.
- Arm B: Topical Naltrexone Cream (Experimental): Patients will start with placebo in week 2 and move on to naltrexone treatment in week 3. There will be a wash-in phase during week 1. Following week 2 and week 3, at visits 3 and 4, patients will be asked for the area where they are experiencing most intense itch and the investigators will take suction blisters from that area before any treatment. They will be told to bring the medication they have been using and they will apply this topically. After an hour, another suction blister will be taken from the same area. This will ensure the study is still blinded as neither the physician or the participant will know whether the medication was a placebo or not. Participants may apply their topical treatment as often as he wishes.
  Interventions: Drug: Naltrexone
- Arm C: Placebo Cream (Placebo Comparator): Patients will start with naltrexone treatment in week 2 and move on to placebo treatment in week 3. Other than this, all procedures will be the same as in study arm B.
  Interventions: Other: Placebo Cream

INTERVENTIONS:
Drug: Naltrexone — Topical naltrexone cream (1%)
  Arms: Arm B: Topical Naltrexone Cream
Other: Placebo Cream — Topical placebo cream
  Arms: Arm C: Placebo Cream

SUMMARY:
To study the etiology and the epigenetic pathways leading to and regulating chronic itch. Similarly, to examine the mechanisms underlying skin changes, including epigenetic alterations while also testing the efficacy of medications, especially topical intervention. In this study, the investigators aim to examine chronic sensory disorder mechanisms related to chronic itch.

DETAILED DESCRIPTION:
Itch was recently identified as one of the top three priority topics in dermatology at a Research Agenda Conference sponsored by the American Academy of Dermatology in 2012. Chronic itch is a complex phenomenon, involving the skin, immune and nervous systems to various degrees. Therefore, focusing on a particular pruritic disease will enable us to work out the underlying pathophysiological mechanisms that occur between the skin and the brain to establish a rational treatment approach.

Atopic Dermatitis (AD) is defined as a chronic inflammatory dermatological disease characterized by immunological and neurological cutaneous hyperreactivity with ongoing itch and inflammation. It is linked to an atopic predisposition with skin barrier abnormalities, recurrent delayed-type inflammations; frequently the development of IgE-mediated inhalant and gastrointestinal-related immediate type reactions. It is estimated that the prevalence for AD is at least 17% of the population lifetime worldwide with some reports of increasing prevalence in the last decades. It is also increasingly being observed in the aging population with dry, itchy skin.

Various topical and systemic therapies are available and choices are based on disease extent, presence of acute flare, and age of the patient. Unfortunately, itch in AD can be challenging to control; although multiple topical and systemic treatments are available, to date no universally accepted treatment exists.

The investigators have previously shown that opioid receptors play an important role in pruritus. Therefore, the investigators plan on expanding on previous and ongoing experiences with opioid antagonists and study the epigenetic and molecular mechanisms behind. Moreover, the investigators have recently discovered that the endogenous opioid ligand Met-Enkephalin influences circadian rhythm by binding directly to CLOCK gene promoters in the nucleus, which then change the amplitude and phase-shift these genes in keratinocytes.

Ultimately, the investigators would like to evaluate the effectiveness of topical application of Naltrexone in an effort to potentially help to treat chronic, untreatable itch and learn more about peripheral disorders of sensation (itch and pain).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD via simplified UK Working Group Criteria and a baseline PSGA score of 2 or greater
* Subjects taking hormone-containing medications must be on a stable dose for 6 months prior to study start to avoid any confounding influence on sensory and pain perception

Exclusion Criteria:

* Use of topical or oral anti-inflammatory medications for 2 weeks prior to the study start
* Use of topical or oral anti-histamines for 2 weeks prior to the study start
* Use of topical or oral anti-pruritic agents for 2 weeks prior to the study start
* Use of oral neuromodulatory agents for 2 months prior to study start
* Current use of chronic pain medications (including opioids, antidepressants and anti-epileptic drugs)
* Use of nicotine-containing products for the past 6 months prior to study start
* History of radiation or chemotherapy
* History of traumatic injury on prospective test sites
* Unstable thyroid function within the past 6 months prior to study start to exclude thyroid-related neuropathy (Duyff et al, 2000)
* Known history of central or peripheral nervous system dysfunction
* History of acute hepatitis, chronic liver disease or end stage liver disease
* History of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome
* History of neuropathy associated with chronic obstructive pulmonary disease, diabetes mellitus, documented exposure to organophosphates or heavy metals or polychlorinated biphenyls
* Known nutritional deficiency (vitamin B12, vitamin D, iron or zinc) within 3 months prior to the study start
* Use of illicit drugs within the past 6 months prior to study start
* History of daily use of power tools
* Lyme disease, porphyria, rheumatoid arthritis, Hansen's disease (leprosy) or use of antineoplastic chemotherapeutic agents
* Subject has any medical condition that, in the judgment of the Investigator, would jeopardize the subject's safety following exposure to the administered medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for Itching: Circadian 2 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+2h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Circadian 4 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+4h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Circadian 6 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+6h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Circadian 8 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+8h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Circadian 10 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+10h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Circadian 12 Hours AW | 7 days
  To assess the effects of circadian rhythm on pruritus, participants will record itch intensity using a visual analog scale (VAS) at the following time points after waking (AW): AW+12h for 7 days. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) of 7 daily measurements will be reported.
Visual Analog Scale for Itching: Treatment 0 min | 0 minutes after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 0 minutes after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 20 min | 20 minutes after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 20 minutes after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 40 min | 40 minutes after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 40 minutes after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 1 Hour | 1 hour after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 1 hour after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 2 Hours | 2 hours after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 2 hours after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 3 Hours | 3 hours after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 3 hours after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.
Visual Analog Scale for Itching: Treatment 4 Hours | 4 hours after applying topical cream
  To assess the effects of naltrexone 1% or placebo cream on pruritus, participants will record itch intensity using a visual analog scale (VAS) at 4 hours after applying cream for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). The mean (in millimeters) over 3 pruritis attacks will be reported.

SECONDARY OUTCOMES:
Time to Itching Intensity Decrease by 50% | 4 hours
  Time to itching intensity decrease by 50% using visual analog scale (VAS) after applying topical cream (either naltrexone or placebo) for 3 pruritis attacks in 1 week. VAS ranges from 0mm (no itch) to 100mm (unbearable itch). VAS will be recorded at 6 time points after application (AA) of cream: 0minAA, 20minAA, 40minAA, 60minAA, 120minAA, 180minAA, and 240minAA. The mean value (in min AA) across 3 pruritis attacks in 1 week will be reported.
Total Reduction in Itch Intensity | 4 hours
  The total reduction of itch intensity as measured by visual analog scale (VAS) after applying topical cream (either naltrexone or placebo). VAS ranges from 0mm (no itch) to 100mm (unbearable itch). Participants will measure itching via VAS at 0min after cream application and 4hr after cream application. Total reduction in itch will be measured in millimeters on VAS. The mean value (across 3 pruritis attacks in 1 week) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bigliardi, MD, Principal Investigator — University of Minenesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No